CLINICAL TRIAL: NCT04755465
Title: Effects of Neuromuscular Electrical Stimulation Combined With Resistance Exercises on Muscle Strength in Adult Hematological Cancer Patients: A Randomized Controlled Study
Brief Title: Effects of NMES and Exercise in Hematological Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Elif Esma Safran, Lecturer, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-16/10
Record Dates: First submitted 2021-02-07; First posted 2021-02-16 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Hematologic Malignancy; Muscle Weakness
Keywords: Hematology; Therapeutic Electrical Stimulation; Exercise Therapy
MeSH Terms: conditions — Hematologic Neoplasms; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Exercise Group (Experimental): The lower extremity resistance exercise (REx) program was designed by reviewing the exercise principles recommended by the ACSM and the literature on physical activity and hematological cancer patients. The patients were treated for 40-60mins, 6 weeks. The exercise program includes active movements of the upper and lower extremities, stretching exercises, and resistance exercises for the lower extremities. REx to be applied with resistance bands of different resistance or with the patient's body weight. Clinical force generation of therapy bands follows a progression. Our proposed training protocol includes 4-6 different exercises for each extremity. Intensity, sets, and reps were adjusted to a target score of 12 to 14 using the Borg scale. Patients performed 1 set of 10 repetitions of each REx based on their fatigue level. Intensity (~ RPE 15-16) and resistance were gradually increased. When the patient complained of extreme fatigue, the resistance was reduced to the previous level.
  Interventions: Other: Structured Exercise
- NMES Training Group (Experimental): In addition to resistance exercises, NMES will be applied to the quadriceps muscles in both legs of the patients in this group. The application will be made with a portable device using disposable electrodes. One of the electrodes will be placed proximally, that is, at the midpoint of the quadriceps muscle, while the second electrode will be placed on the distal part. In order to ensure that the patients get used to the device, low-intensity current with a frequency range of 5 Hz, 10-30 minutes. Afterward, the treatment program will continue with a high-frequency current with a frequency range of 50 Hz, 15 minutes. Participants were instructed to voluntarily contract the quadriceps muscles during periods of HF-NMES stimulation to increase the strengthening effect and improve NMES tolerance.
  Interventions: Device: Neuromuscular Electrical Stimulation; Other: Structured Exercise

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Neuromuscular Electrical Stimulation (NMES) is based on the principle of creating a contraction by stimulating the nerve fibers innervating the related muscle in the healthy muscle and the muscle fibers in the denervated muscle with electrical current. The electric currents used in stimulation of muscles and nerves perform this function by changing the electrical potential of cell membranes.
  It is contraindicated in pregnancy, presence of pacemaker, severe heart disease, epilepsy, fracture, dementia and impaired consciousness. We prevent contraindicated situations by excluding volunteer participants with these characteristics.
  Arms: NMES Training Group
Other: Structured Exercise — Warm-up exercise, main training program and cool down exercise. Main training consists of resistance exercises to be applied with resistance bands of different resistance or with the patient's own body weight. Our prescribed training protocol includes 4-6 different exercises for each limb (bench press with resistance band, upper extremity proprioceptive neuromuscular facilitation exercises, biceps/triceps curl, leg press, knee extension, 4-way hip motion, mini squat). Intensity, sets, and number of repetitions will be adapted to a target score between 12 and 14 using the Borg scale. It will be applied as low intensity, long-term passive stretching exercises to the pectoral, hamstring, and gastrosoleus muscle groups. Patients will perform 1 set of 10 repetitions of each resistance exercise determined by their level of fatigue. Resistance will be increased every three visits. If the patient complains of excessive fatigue, the resistance will be reduced to the previous level.

SUMMARY:
Physical activity levels of adult hematologic cancer patients are deficient. The resulting physical inactivity causes fatigue, muscle loss, and deterioration in physical performance values. However, physical exercise programs still play a minor role in treating hematological malignancies. In addition, there are no reliable data in the literature regarding risk factors, feasibility, and exercise results in individuals with hematological malignancies. Although it is known that the use of corticosteroids, which are among the drugs given during chemotherapy, causes muscle weakness, there are no physical exercise programs performed with this patient group in the literature. The current study aims to compare the effects of resistance exercise and resistance exercise combined with neuromuscular electrical stimulation on muscle strength, functional lower extremity strength, and mobility in hematological cancer patients during chemotherapy.

DETAILED DESCRIPTION:
Although people with hematological malignancies have to endure long stages of treatment and inactivity that are known to reduce their physical performance levels, it is still common practice to rest and avoid intense exercise. Although physical activity and exercise are important approaches to many diseases, their effects on cancer have been studied recently. There are still not enough studies in this area and it is not widely used. In recent studies, it is thought that exercise may benefit the symptoms that develop due to treatment in cancer patients. Even in the presence of severe muscle weakness and fatigue, skeletal muscle provides great adaptation when there is an appropriate exercise stimulus. In addition, exercise can increase immune functions, so it is thought that exercise practices in hematological cancer patients can specifically improve cellular functions such as microbial phagocytosis, T-cell proliferation, vaccine response, and killing tumor cells. There are various studies and approaches that try to create a different strategy and include physical exercise in the treatment strategy of hematological malignancies. These exercise programs generally include aerobics, flexibility, and resistance training methods. The necessity of developing alternative methods to exercise is emphasized in the literature due to the development of complications that affect participation in basic exercises such as walking. Resistance exercise training has been effective in improving muscle strength and endurance in cancer survivors, with most of the research on those with breast cancer, prostate cancer, and head and neck cancer. The number of studies providing strengthening training in patients with hematological cancer is limited. Neuromuscular electrical stimulation (NMES) has proven efficacy in improving muscle strength in a variety of populations. NMES training also has applicability for the cancer population to prevent treatment-related complications and improve health-related quality of life. However, there is still no high-level evidence to support the administration of NMES in cancer patients. In the present study, we aimed to evaluate the effect of resistance exercise improve muscle weakness in hematological cancer patients receiving intensive chemotherapy after HSCT. In addition, we aimed to evaluate the effect of resistance exercise and NMES training on fatigue, mobility, and quality of life in hematological cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hematological cancer,
* ≥ 18 years old
* ECOG Performance Status to be between 1-3
* Hemoglobin; 8-10gr / dl and over
* Receiving platelet support related to thrombocytopenia and/or having a platelet value of 20.000 mm3 or more
* Leukocyte (WBC) count being 3000 μL and above
* Giving written consent to participate in the study

Exclusion Criteria:

* Comorbidities that cause fatigue (eg multiple sclerosis, Parkinson's disease, heart failure)
* Presence of previously diagnosed heart disease
* Using a pacemaker
* Rapid deterioration of the general condition (sudden uncontrolled weight loss, confused consciousness, high C reactive protein (CRP) values)
* Brain metastasis or femoral bone metastasis
* Having dementia or psychotic condition
* Being depressed and /or taking medication to treat depression
* Presence of epilepsy
* Presence of neuropathy
* Having sensory defects in the NMES application area
* Denying NMES application

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Evaluation | Change from Baseline Muscle Strength through study completion, an average of 6 weeks
  Participants' muscle strength measurements will be made using a digital hand dynamometer (J Tech Commander Muscle Tester). The patients will be seated in the appropriate position and the dynamometer will be placed in the dominant leg to give resistance to the muscle to be evaluated. While patients press the dynamometer as hard as possible for three seconds, the evaluator will give resistance to prevent any movement to provide an isometric contraction. Following the familiarization test, patients will perform three trials with standardized verbal encouragement and the highest strength (kilogram, kg) sustained for over half a second will be recorded.
Functional Muscle Strength Evaluation | Change from Baseline Functional Muscle Strength through study completion, an average of 6 weeks
  Lower extremity functional strength will be evaluated using the "Sit and Stand for 30 sec" test. The patient will be instructed to stand up and sit back and forth from a standardized chair as quickly as possible in 30 seconds without using his arms. Participants will be able to use their hands to help them stand as needed, and standardized verbal encouragement will be provided to continue sitting and standing throughout the test.

SECONDARY OUTCOMES:
Anthropometric Assessment | Baseline and Immediately after completion of study, an average of 6 weeks
  Thigh circumference measurement will be made from the middle of the thigh over the Quadriceps muscle. By marking the inguinal region and the proximal part of the patella, the midpoint between the two points will be found. All measurements will be made on the right side and by the same physiotherapist.
Mobility Assessment | Baseline and Immediately after completion of study, an average of 6 weeks
  "Timed Up-Go Test" will be applied before and after treatment to evaluate the patient's mobility and functional exercise capacity. The time taken to complete the task is strongly correlated with the level of functional mobility. In other words, the longer the person completes the task, the more dependent he is on daily life activities.
The Brief Fatigue Scale | Baseline and Immediately after completion of study, an average of 6 weeks
  The Brief Fatigue Scale will be used to assess cancer-related fatigue in our study. This scale is one of the standard tests used to evaluate fatigue in cancer patients. Evaluates the level of fatigue in the last 24 hours and the effect of fatigue on daily activities (general activity, mood, walking ability, work life, relationships with other people, joy of life)
European Cancer Research and Treatment Organization Quality of Life Questionnaire | Baseline and Immediately after completion of study, an average of 6 weeks
  The assessment of quality of life will be carried out using the European Cancer Research and Treatment Organization Quality of Life Questionnaire Version 3.0. The scale consists of three subsections: general health status scale, functional scale, and symptom scale, and includes a total of 30 questions.

OTHER OUTCOMES:
Eastern Cooperative Oncology Group Performance Status Scale | Baseline and Immediately after completion of study, an average of 6 weeks
  An overall assessment of activity level will be based on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale based on the degree of muscle weakness found in the Cancer Treatment Evaluation Program Common Toxicity Criteria, and patients with an ECOG performance status of 1-3 will be treated.

CONTACTS AND LOCATIONS:
Overall Officials: Ant Uzay, MD, Study Director — Acibadem Healthcare Group; Fatma Mutluay, Prof, Study Director — Medipol University; Elif Es Safran, MSc, Principal Investigator — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After completion of study

REFERENCES:
- [Derived] Safran EE, Mutluay F, Uzay A. Effects of neuromuscular electrical stimulation combined with resistance exercises on muscle strength in adult hematological cancer patients: A randomized controlled study. Leuk Res. 2022 Oct;121:106932. doi: 10.1016/j.leukres.2022.106932. Epub 2022 Aug 22. PMID 36027848